CLINICAL TRIAL: NCT05604170
Title: A Phase 3, Open-label Study of Adjunctive Ganaxolone (GNX) Treatment in Children and Adults With Tuberous Sclerosis Complex (TSC)-Related Epilepsy (TrustTSC OLE)
Brief Title: Open-label Study of Adjunctive GNX Treatment in Children and Adults With TSC-related Epilepsy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1042-TSC-3002
Record Dates: First submitted 2022-10-05; First posted 2022-11-03 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Tuberous Sclerosis Complex
Keywords: Tuberous Sclerosis Complex-Related Epilepsy; Ganaxolone; Adjunctive
MeSH Terms: conditions — Tuberous Sclerosis | interventions — ganaxolone

STUDY DESIGN:
Masking Description: This is an open-label, single arm study with no blinding as all participants will receive adjunctive GNX
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ganaxolone (GNX) oral suspension, 3 times a day (TID) (Experimental)
  Interventions: Drug: Ganaxolone

INTERVENTIONS:
Drug: Ganaxolone — GNX will be administered.

SUMMARY:
This is a Phase 3, global, open-label extension (OLE) study of adjunctive GNX treatment in children and adults with TSC who previously participated in either Study 1042-TSC-3001 or Study 1042-TSC-2001

ELIGIBILITY:
Inclusion Criteria:

1. Completion of Study 1042-TSC-3001 or participants who continue to meet study requirements in Study 1042-TSC-2001.
2. Participant/parent(s)/LAR(s) willing and able to give written informed consent/assent, after being properly informed of the nature and risks of the study and prior to engaging in any study-related procedures. If the participant is not qualified or able to provide written informed consent based on age, developmental stage, intellectual capacity, or other factors, parent(s)/LAR(s) must provide assent for study participation, if appropriate.
3. Parent(s)/caregiver(s) is (are) willing and able to maintain an accurate and complete daily seizure diary for the duration of the study.
4. Willing and able to take Investigational product (IP) (suspension) as directed with food TID.
5. Women of childbearing potential (WOCBP) must be using a medically acceptable method of birth control and have a negative quantitative serum beta-human chorionic growth hormone (β-HCG) test collected at the initial visit. Childbearing potential is defined as a female who is biologically capable of becoming pregnant. Medically acceptable methods of birth control include intrauterine devices (that have been in place for at least 1 month prior to the screening visit), hormonal contraceptives (eg, combined oral contraceptives, patch, vaginal ring, injectables, and implants), and surgical sterilization (such as oophorectomy or tubal ligation). When used consistently and correctly, "double-barrier" methods of contraception can be used as an effective alternative to highly effective contraception methods. Contraceptive measures such as Plan B™, sold for emergency use after unprotected sex, are not acceptable methods for routine use
6. Male participants must agree to use highly effective contraceptive methods during the study and for 30 days after the last dose of IP. Highly effective methods of contraception include surgical sterilization (such as a vasectomy) and adequate "double-barrier" methods.

Exclusion Criteria:

1. Pregnant or breastfeeding.
2. An active Central nervous system (CNS) infection, demyelinating disease, or degenerative neurological disease.
3. History of psychogenic nonepileptic seizures.
4. Any disease or condition (other than TSC) at the initial visit that could compromise the hematologic, cardiovascular (including any cardiac conduction defect), pulmonary, renal, gastrointestinal, or hepatic systems; or other conditions that might interfere with the absorption, distribution, metabolism, or excretion of the IP, or would place the participant at increased risk or interfere with the assessment of safety/efficacy. This may include any illness in the past 4 weeks which in the opinion of the investigator may affect seizure frequency.
5. Unwillingness to avoid excessive alcohol use or cannabis use throughout the study.
6. Have active suicidal plan/intent or have had active suicidal thoughts in the past 6 months or a suicide attempt in the past 6 months.
7. Known sensitivity or allergy to any component in the IP(s), progesterone, or other related steroid compounds.
8. Exposed to any other investigational drug (except for GNX in Study 1042-TSC-2001 or Study 1042-TSC-3001) or investigational device within 30 days or fewer than 5 half-lives prior to Visit 1 (first visit of the OLE). For therapies in which half-life cannot be readily established, the Sponsor's medical monitor should be consulted.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (20):
  - Arkansas Children's Research Institute, Little Rock, Arkansas
  - UCLA Mattel Children's Hospital, TSC Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Hospital - Delaware Valley, Wilmington, Delaware
  - Boston Children's Hospital, Harvard Medical School, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health/Levine Children's Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Child Neurology Consultants of Austin (CNCA), Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - McGovern Medical School at the University of Texas Health Science Center, Houston, Texas
  - University of Utah Health Care-Pediatric Neurology, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Australia (4):
  - Austin Health, Heidelberg
  - Royal Brisbane and Women's Hospital, Herston
  - Alfred Health, Melbourne
  - Royal Melbourne Hospital, Parkville
- Canada (5):
  - Hôtel Dieu de Montréal - CHUM, Montreal
  - CHU Sainte-Justine, Montreal
  - The Hospital for Sick Children, Toronto
  - Toronto Western Hospital, Toronto
  - BC Children's Hospital, Vancouver
- China (5):
  - Peking University First Hospital, Beijing
  - Beijing Children Hospital, Capital Medical University, Beijing
  - Chinese PLA General Hospital, Beijing
  - The Affiliated Hospital of Guizhou Medical University, Beijing
  - First Hospital of Jilin University, Jilin
- France (3):
  - University Hospital of Lyon, Bron
  - Hôpital Sud, Rennes
  - University of Strasbourg, Strasbourg
- Germany (6):
  - Epilepsie-Zentrum Bethel - Krankenhaus Mara, Bielefeld
  - University Hospital Bonn, Bonn
  - ZNN - Epilepsiezentrum Frankfurt am Main, Frankfurt
  - Universitäts Krankenhaus Freiburg, Freiburg im Breisgau
  - Gemeinschaftskrankenhaus Herdecke, Herdecke
  - Epilepsiezentrum Kleinwachau gGmbH, Radeberg
- Schneider Children´s Medical Center, Petah Tikva, Israel
- Italy (2):
  - Pediatric Neurology and Muscular Diseases Unit - University of Genoa, Genova
  - Policlinico Umberto I, Rome
- Spain (6):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Ruber International, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario y Politécnico La Fe, Valencia
- United Kingdom (2):
  - Bristol Royal Hospital for Children, Bristol
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total 117 participants entered the OLE phase and had received at least 1 dose of Ganaxolone (GNX). Of these 8 were previously in Study 1042-TCS-2001 and 109 were previously in Study 1042-TCS-3001 and met eligibility criteria for continued treatment.
Pre-assignment Details: Participants who completed Study 1042-TCS-2001 and 1042-TCS-3001 were enrolled in the Open-Label Extension (OLE) phase and the study was terminated prematurely due to Sponsor decision.
Groups:
- Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID): Participants received 50 mg/mL oral suspension containing 110 mL Ganaxolone (GNX), 3 times a day (TID) with food.
Period: Overall Study
Arm/Group | Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID)
Started | 117
Completed | 0
Not Completed | 117
Not completed — Lack of Efficacy | 5
Not completed — Adverse Event | 6
Not completed — Physician Decision | 6
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 11
Not completed — Early study termination by sponsor | 77
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Population: Safety analysis set comprised of all participants who received at least 1 dose of the investigational product (IP).
Arm/Group | Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID)
Number analyzed (Participants) | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 24
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 82
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Treatment Emergent Adverse Events (TEAEs), Serious TEAEs and Withdrawals and Dose-Reductions Due to AEs
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study patient, temporally associated with the use of study drug, whether or not considered related to the study drug. A serious adverse event was any untoward medical occurrence that, at any dose, results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or any other event that requires scientific judgment.
Time Frame: Up to 150 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID)
Number analyzed (Participants) | 117
Participants
  Any serious TEAE | 21
  Any TEAE | 79
  Withdrawals Due to AEs | 6
  Dose-Reduction Due to AEs | 16

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Parameters
Description: Vital parameters including heart rate, respiration rate, blood pressure, and body temperature were measured in seated position for at least 5 minutes.
Time Frame: Up to 150 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID)
Number analyzed (Participants) | 117
Participants | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Physical Examinations
Description: Physical examinations included a full physical evaluation of body systems including: General appearance, head (eyes, ears, nose, and throat), cardiovascular, respiratory, gastrointestinal, genitourinary, musculoskeletal, endocrine/metabolic, hematologic/lymphatic, skin, and other systems as appropriate.
Time Frame: Up to 150 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID)
Number analyzed (Participants) | 117
Participants | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Neurological Examinations
Description: Neurological examinations included an evaluation of: Cranial nerves, motor exam, sensory exam, reflexes, coordination/cerebellar
Time Frame: Up to 150 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID)
Number analyzed (Participants) | 117
Participants | 0

5. Primary Outcome: Number of Participants With Clinically Significant Changes in Developmental Examinations
Description: Developmental examinations (applicable only to pediatric participants 1 to 17 years of age, inclusive) included an evaluation of speech/language, motor skills, and social skills
Time Frame: Up to 150 Weeks
Population: Safety Analysis Set. Only pediatric participants of 1 to 17 years of age were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID)
Number analyzed (Participants) | 72
Participants | 0

6. Primary Outcome: Number of Participants With Clinically Significant 12-lead Electrocardiogram (ECG) Findings
Description: Twelve-lead ECGs were performed by the physician using an ECG machine that automatically calculates the heart rate and measure PR, QRS, QT and QTc intervals.
Time Frame: Up to 150 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID)
Number analyzed (Participants) | 117
Participants | 0

7. Primary Outcome: Number of Participants With Clinically Significant Changes in Hematology Parameters
Description: Blood samples were collected for the analysis of hematology parameters: hemoglobin, hematocrit, erythrocytes, thrombocytes (platelet count). Differential blood counts, including basophils, eosinophils, neutrophils, lymphocytes, and monocytes
Time Frame: Week 1 through Week 150
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID)
Number analyzed (Participants) | 117
Participants | 0

8. Primary Outcome: Number of Participants With Clinically Significant Changes in Chemistry Parameters
Description: Blood samples were collected for the analysis of chemistry parameters: blood urea nitrogen (BUN), potassium, alanine aminotransferase (ALT), alkaline phosphatase (ALP)/serum glutamic pyruvic transaminase (SGPT), total bilirubin, creatinine, sodium, aspartate aminotransferase (AST)/serum glutamic oxaloacetic (SGOT), total protein, fasting blood glucose, calcium, carbon dioxide, estimated glomerular filtration rate (eGFR), and chloride
Time Frame: Up to 150 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID)
Number analyzed (Participants) | 117
Participants | 0

9. Primary Outcome: Number of Participants With Clinically Significant Changes in Urinalysis
Description: Urine samples were collected for the analysis of urinalysis parameters: Specific gravity, color, clarity, pH, glucose, protein, blood, nitrite, protein, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase by dipstick, and microscopic examination (if blood or protein was abnormal)
Time Frame: Up to 150 Weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID)
Number analyzed (Participants) | 117
Participants | 0

10. Primary Outcome: Number of Participants (Age Greater Than 17 Years) With Abnormal Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a clinician administered assessment tool that evaluates suicidal ideation and behavior. Number of participants that have an affirmative response to the 5 items for suicidal ideation (1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation with any methods (not plan) without intent to act, 4. Active suicidal ideation with some intent to act, without specific plan, 5. Active suicidal ideation with specific plan and intent) and/or to the 5 items for suicidal behavior (1. Preparatory acts or behavior, 2. Aborted attempt, 3. Interrupted attempt, 4. Actual attempt, 5. Completed suicide) will be reported. The score ranges from 1 to 5 and higher scores indicate worse symptoms.
Time Frame: Up to Week 52
Population: Safety Analysis Set. Only those participants with data available at specified timepoints have been analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID)
Number analyzed (Participants) | 45
Participants
  Suicidal Behavior: Preparatory acts or behavior | 0
  Suicidal Behavior: Aborted attempt | 0
  Suicidal Behavior: Interrupted attempt | 0
  Suicidal Behavior: Actual attempt | 0
  Suicidal Behavior: Completed suicide | 0
  Suicidal Ideation: Wish to be dead | 0
  Suicidal Ideation: Non-specific Active thoughts | 0
  Suicidal Ideation: Active ideation without intention to act | 0
  Suicidal Ideation: Active ideation with some intent to act without a plan | 0
  Suicidal Ideation: Active ideation with a specific plan and intent | 0
  Non-suicidal Self-Injurious Behavior | 1

11. Secondary Outcome: Percent Change From Baseline in 28-day Seizure Frequency During Open Label Extension
Description: Seizure frequency will be calculated as the total number of seizures divided by the number of days with seizure data, multiplied by 28. Percent change from baseline in 28-day frequency was calculated for each participant by subtracting Baseline 28-day seizure frequency from post-Baseline 28-day seizure frequency, whole divided by Baseline 28-day seizure frequency and multiplied by 100.
Time Frame: Baseline (Day 1), Week 52
Population: Intent to Treat comprised all participants who received at least 1 dose of the IP. Only those participants with data available at specified timepoints have been analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID)
Number analyzed (Participants) | 107
percent change | -31.59 (113.997)

ADVERSE EVENTS:
Time Frame: Up to 150 Weeks
Description: Serious TEAEs and TEAEs were collected in the Safety Analysis Set which comprised of all participants who received at least 1 dose of the investigational drug.
Arm/Group | Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID)
All-Cause Mortality (participants affected / at risk) | 1/117
Serious Adverse Events (participants affected / at risk) | 21/117
Other Adverse Events (participants affected / at risk) | 79/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID) (N=117)
Pneumonia (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 2
Atypical Pneumonia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Covid-19 (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Pneumonia Bacterial (Infections and infestations) | 1
Pneumonia Mycoplasmal (Infections and infestations) | 1
Respiratory Syncytial Virus Infection (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 1
Seizure (Nervous system disorders) | 5
Status Epilepticus (Nervous system disorders) | 1
Pyrexia (General disorders) | 1
Sudden Unexplained Death In Epilepsy (General disorders) | 1
Inappropriate Affect (Psychiatric disorders) | 1
Mental Status Changes (Psychiatric disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Embedded Device (Product Issues) | 1
Urethral Haemorrhage (Renal and urinary disorders) | 1
Urethral Prolapse (Renal and urinary disorders) | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (GNX) Oral Suspension, 3 Times a Day (TID) (N=117)
Upper Respiratory Tract Infection (Infections and infestations) | 10
Pneumonia (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 7
Covid-19 (Infections and infestations) | 4
Ear Infection (Infections and infestations) | 4
Influenza (Infections and infestations) | 3
Pharyngitis Streptococcal (Infections and infestations) | 3
Urinary Tract Infection (Infections and infestations) | 3
Gastroenteritis Viral (Infections and infestations) | 2
Respiratory Syncytial Virus Infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 2
Acarodermatitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Gastroenteritis Bacillus (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Kidney Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Viral Infection (Infections and infestations) | 1
Viral Myositis (Infections and infestations) | 1
Seizure (Nervous system disorders) | 17
Somnolence (Nervous system disorders) | 10
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Sedation (Nervous system disorders) | 2
Status Epilepticus (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Drooling (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Parkinsonism (Nervous system disorders) | 1
Psychomotor Hyperactivity (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Aphthous Ulcer (Gastrointestinal disorders) | 1
Dental Caries (Gastrointestinal disorders) | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 1
Mouth Ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Salivary Hypersecretion (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 9
Fatigue (General disorders) | 5
Decreased Activity (General disorders) | 1
Pain (General disorders) | 1
Swelling (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 6
Foot Fracture (Injury, poisoning and procedural complications) | 2
Ligament Sprain (Injury, poisoning and procedural complications) | 2
Clavicle Fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Face Injury (Injury, poisoning and procedural complications) | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1
Hand Fracture (Injury, poisoning and procedural complications) | 1
Ligament Rupture (Injury, poisoning and procedural complications) | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1
Periorbital Haematoma (Injury, poisoning and procedural complications) | 1
Skin Laceration (Injury, poisoning and procedural complications) | 1
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1
Tooth Fracture (Injury, poisoning and procedural complications) | 1
Sleep Disorder (Psychiatric disorders) | 3
Abnormal Behaviour (Psychiatric disorders) | 2
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Confusional State (Psychiatric disorders) | 1
Irritability (Psychiatric disorders) | 1
Suicidal Ideation (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2
Abnormal Weight Gain (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Dyshidrotic Eczema (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Shagreen Skin (Skin and subcutaneous tissue disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 3
Amenorrhoea (Reproductive system and breast disorders) | 1
Menstrual Disorder (Reproductive system and breast disorders) | 1
Menstruation Irregular (Reproductive system and breast disorders) | 1
Weight Increased (Investigations) | 2
Blood Homocysteine Increased (Investigations) | 1
Electrocardiogram Abnormal (Investigations) | 1
Electrocardiogram Qt Prolonged (Investigations) | 1
Specific Gravity Urine Increased (Investigations) | 1
Bundle Branch Block Right (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal Pain (Renal and urinary disorders) | 1
Haematoma (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Chalazion (Eye disorders) | 1
Scleral Discolouration (Eye disorders) | 1
Allergy To Arthropod Bite (Immune system disorders) | 1
Seasonal Allergy (Immune system disorders) | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Angiofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fibrous Histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Central Hypothyroidism (Endocrine disorders) | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 1
Hepatic Lesion (Hepatobiliary disorders) | 1
Mastoiditis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT05604170/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT05604170/SAP_002.pdf